CLINICAL TRIAL: NCT01622270
Title: Energy Expenditure in Patients With Crohn's Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-12-NV-533-CTIL
Record Dates: First submitted 2012-06-05; First posted 2012-06-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-01

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Calorimetry, Indirect; Body Composition

STUDY DESIGN:
Observational Model: Case-Only

INTERVENTIONS:
Other: Indirect calorimetry, body composition , blood tests,3 days food records,Crohns disease activity index — Indirect calorimetry test by a indirect calorimeter (OHMEDA) body composition by a DEXA machine blood tests, 3 days food records, Crohns disease activity index

SUMMARY:
The objective of this study is to investigate the changes in crohn on resting energy expenditure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohn's disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with Crohn's disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
changes in crohn on resting energy expenditure | two weeks